CLINICAL TRIAL: NCT03920956
Title: Implementation & Evaluation of a 24-Hour Ambulatory Blood Pressure Monitoring Service in Community Pharmacies
Brief Title: 24-Hour Ambulatory Blood Pressure Monitoring in Community Pharmacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HM20015789
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 24-hour ABPM by Pharmacists (Experimental): Patients will meet with the pharmacist to be equipped with a 24-hour ambulatory blood pressure monitor (ABPM). Patients will return the monitor for the pharmacists to download the results to send to their medical provider.
  Interventions: Other: ABPM service by Pharmacists

INTERVENTIONS:
Other: ABPM service by Pharmacists — Patients will receive ABPM services provided by a pharmacist and complete a patient satisfaction survey

SUMMARY:
This study is designed to explore the feasibility of providing 24-hour ambulatory blood pressure monitoring in community pharmacies. The investigators hypothesize it will be feasible for community pharmacies to provide the service to assist medical providers in the diagnosing and management of high blood pressure. The investigators will also survey participants regarding their experience with the service as well as conduct interviews with participating pharmacists and medical providers to understand their views and opinions on the feasibility of the service.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years of age suspected by their physician of having "white coat" or "masked" hypertension (HTN), hypotension symptoms due to antihypertensive therapy, uncontrolled sustained HTN, requiring additional confirmation of an initial diagnosis if HTN, or resistant HTN.

Exclusion Criteria:

* Documented past medical history of persistent atrial fibrillation, on hemodialysis, pregnancy, or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with the pharmacy service and experience wearing the ABPM | up to 72 hours
  Patient satisfaction will be assessed using a 9 item survey. Participants will rate items on a 5-point scale from strongly agree to strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Dixon, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khaddage SJ, Patterson JA, Sargent LJ, Price ET, Dixon DL. Sex and Age Differences in Ambulatory Blood Pressure Monitoring Tolerability. Am J Hypertens. 2021 Apr 20;34(4):335-338. doi: 10.1093/ajh/hpaa182. PMID 33180905